CLINICAL TRIAL: NCT06597136
Title: Examination of the Effects of Kinesiology Tape Application for Respiratory Muscles on Early Functional Level and Respiratory Function in Intensive Care Unit Patients
Brief Title: The Effect of Kinesiology Tape Application on Functional Level and Respiratory Function in Intensive Care Unit Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istinye University (Other)
Responsible Party: Principal Investigator, Yasemin Çırak, Principal Investigator, Istinye University
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Supportive Care
Other Study IDs: IstinyeU-ORSELOGLU-001
Record Dates: First submitted 2024-05-01; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: İntensive Care Patients
Keywords: intensive care; respiratory muscle strength; respiratory function; kinesiotape
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: In the 1st group, only conventional treatment will be applied, in the 2nd group, diaphragmatic kinesiology taping will be applied in addition to conventional treatment, in the 3rd group, kinesiological taping will be applied to the auxiliary respiratory muscles in addition to conventional treatment, and in the 4th group, sham taping will be applied.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Diaphragmatic kinesiology taping (Experimental): The taping on the diaphragm from the abdomen was performed when the participant was standing and breathed-out and the body was in extension. The base of the tape was about 1 inch below the xiphoid process area. Then the arms were lifted above the head and, with maximum deep inspiration and after maximum rib cage expansion, the tails were applied with 10% tension on the rib cage. Diaphragmatic kinesiology taping will be applied in addition to conventional treatment for 3 days.
  To evaluate the effectiveness of the application, vital signs, respiratory muscle strength, grip strength, blood gas analysis, dyspnea and fatigue will be evaluated. Additionally, Richmond Agitation Sedation Scale (RASS), Non-Verbal Pain Scale, Glaskow coma scale, Physical Function Test in Intensive Care (PFIT)- CPax (Chelsea Critical Care Physical Assessment Tool) scales will be used.
  Interventions: Other: Diaphragmatic kinesiology taping
- Accessory respiratory muscle kinesiology taping (Experimental): Tapings of the accessory inspiratory muscles were applied in a sitting posture. Sternocleidomastoideus taping was applied when the neck of the participant was in lateral flexion to the opposite side to be taped and in rotation to the same side; and anterior and medius scalene tapings were applied when the neck of the participant was in the lateral flexion position to the opposite side to be taped. Tapings were repeated on the opposite side.Taping was applied to accessory expiratory muscles in the supine position. While the participant was supporting one leg in the hip and knee flexion position on the bed, the other leg was extended from the bed and the hip was kept in the extension position. The obliquus externus muscle was taped on the side with hip-knee flexion and the obliquus internus muscle was taped on the side with hip extension.In addition to conventional treatment, kinesiology taping will be applied to the accessory respiratory muscles for 3 days.
  Interventions: Other: Accessory respiratory muscle kinesiology taping
- Sham kinesiology taping (Sham Comparator): Sham kinesiology taping will be applied for 3 days. Sham KT was performed with the same taping material. A 2-blocked I strip was applied vertically to the sternum. The same procedures were followed.
  To evaluate the effectiveness of the application, vital signs, respiratory muscle strength, grip strength, blood gas analysis, dyspnea and fatigue will be evaluated. Additionally, Richmond Agitation Sedation Scale (RASS), Non-Verbal Pain Scale, Glaskow coma scale, Physical Function Test in Intensive Care (PFIT)- CPax (Chelsea Critical Care Physical Assessment Tool) scales will be used.
  Interventions: Other: Sham kinesiology taping
- Control Group (No Intervention): Conventional treatment will be applied in the control group. Participants' vital signs, respiratory muscle strength, grip strength, blood gas analysis, dyspnea and fatigue will be evaluated. Additionally, Richmond Agitation Sedation Scale (RASS), Non-Verbal Pain Scale, Glaskow coma scale, Physical Function Test in Intensive Care (PFIT)- CPax (Chelsea Critical Care Physical Assessment Tool) scales will be used.

INTERVENTIONS:
Other: Diaphragmatic kinesiology taping — The taping on the diaphragm from the abdomen was performed when the participant was standing and breathed-out and the body was in extension. The base of the tape was about 1 inch below the xiphoid process area. Then the arms were lifted above the head and, with maximum deep inspiration and after maximum rib cage expansion, the tails were applied with 10% tension on the rib cage. Diaphragmatic kinesiology taping will be applied in addition to conventional treatment for 3 days.
  Arms: Diaphragmatic kinesiology taping
Other: Accessory respiratory muscle kinesiology taping — Tapings of the accessory inspiratory muscles were applied in a sitting posture. Sternocleidomastoideus taping was applied when the neck of the participant was in lateral flexion to the opposite side to be taped and in rotation to the same side; and anterior and medius scalene tapings were applied when the neck of the participant was in the lateral flexion position to the opposite side to be taped. Tapings were repeated on the opposite side.Taping was applied to accessory expiratory muscles in the supine position. While the participant was supporting one leg in the hip and knee flexion position on the bed, the other leg was extended from the bed and the hip was kept in the extension position. The obliquus externus muscle was taped on the side with hip-knee flexion and the obliquus internus muscle was taped on the side with hip extension.In addition to conventional treatment, kinesiology taping will be applied to the accessory respiratory muscles for 3 days.
  Arms: Accessory respiratory muscle kinesiology taping
Other: Sham kinesiology taping — Sham kinesiology taping will be applied for 3 days. Sham KT was performed with the same taping material. A 2-blocked I strip was applied vertically to the sternum. The same procedures were followed.
  Arms: Sham kinesiology taping

SUMMARY:
Investigation of the effects of respiratory muscles on the early functional system and respiratory function in the kinesiological period in intensive care patients.

DETAILED DESCRIPTION:
Weakness of respiratory muscles delays weaning from the ventilator, prolongs hospital stay and increases treatment costs. Conventional treatments for respiratory muscles reverse these negative effects. Kinesiology taping has effects that support the muscle to which it is applied, increase circulation and improve its function. Studies have shown positive effects of kinesiology taping applied to COPD patients, and in light of this, it has been predicted that its application to intensive care patients will be beneficial. The results of our study will shed light on the rehabilitation of patients in intensive care and contribute to the literature.

In this study, the investigators aimed to increase the activation of respiratory muscles by taking advantage of the benefits of kinesiology taping in addition to conventional treatment.

Our study, which included a total of 48 participants will consist of 4 groups. Only conventional treatment will be applied to the 1st group, diaphragmatic kinesiology taping will be applied to the 2nd group in addition to conventional treatment, kinesiological taping to the accessory respiratory muscles will be applied to the 3rd group and sham taping will be applied to the 4th group.

ELIGIBILITY:
Inclusion Criteria:

* Individuals receiving inpatient treatment in intensive care who volunteer to participate in the research or who are allowed by their first-degree relatives if they are unconscious,
* Being over 18 years of age
* Being eligible to receive physiotherapy and rehabilitation from an intensive care physician
* Are in clinically stable condition

Exclusion Criteria:

* Patients with coagulation disorders (PT (Prothrombin Time); INR (International Normalized Ratio) value higher than 1.5 and platelet amount less than 50,000 m³)
* Patients with signs of increased intracranial pressure
* Skin wounds, ulcerations, allergic reactions
* Patients in contact isolation due to infection
* In shock
* Having malignancy
* Having multiple organ failure
* Having visual impairment
* Patients who are unconscious

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-09-15 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2024-11-10 (Estimated)

PRIMARY OUTCOMES:
Respiratory Muscle Strength | 3 days
  Maximal inspiratory pressure (MIP) is a measure of the strength of inspiratory muscles, primarily the diaphragm, and allows for the assessment of ventilatory failure, restrictive lung disease and respiratory muscle strength. MIP is measured at residual volume of lung.
Respiratory Muscle Strength | 3 days
  For respiratory muscle strength, maximal expiratory pressure (MEP) will evaluate using an electronic pressure transducer. MEP is measured from total lung capacity.particularly the diaphragm, while MEPs measure the strength of abdominal and intercostal muscles.
  For respiratory muscle strength, maximal inspiratory pressure (MIP), and maximal expiratory pressure (MEP) were evaluated using an electronic pressure transducer. MIP was measured at residual volume, and MEP was measured from total lung capacity
Richmond Agitation-Sedation Scale | 3 days
  Interrater reliability. In many intensive care units, the Richmond Agitation-Sedation Scale(RASS) is used to assess the level of sedation. This scale is designed with a three-step procedure that can help give a RASS score range of -5 to +4.The RASS score ranges from -5 (unarousable) to +4 (combative), with 0 meaning alert and calm.
SOFA (Sequential Organ Failure Assessment) | 3 days
  It evaluates morbidity through six systems (liver, central nervous system, respiratory system, cardiovascular system,renal and coagulation). For each system, points between 1 and 4 are given and the total score is evaluated between 6 and 24. In this score, as the score increases for each system, organ failure is considered to occur.
Visuel Anaolog Scale | 3 days
  A Visual Analogue Scale (VAS) is one of the pain rating scales used for the first time in 1921 by Hayes and Patterson[1]. It is often used in epidemiologic and clinical research to measure the intensity or frequency of various symptoms.For pain intensity according to VAS, "no pain" is usually rated as 0 points and "worst pain imaginable" as 10 points. Ranges for pain intensity; <3. mild pain, 3-6 moderate pain, >6 severe pain
The Glasgow Coma Scale | 3 days
  It is a tool that healthcare providers use to measure decreases in consciousness. The scores from each section of the scale are useful for describing disruptions in nervous system function and also help providers track changes. It's the most widely used tool for measuring comas and decreases in consciousness.The components of the Glasgow Coma Scale include 4 different scores for the eye-opening response, 5 for the verbal response, and 6 for the motor response. The total score has values between 3 and 15. Three is the worst and 15 is the highest.
APACHE II Score | 3 days
  It is a general measure of disease severity based on current physiologic measurements, age & previous health conditions. The score can help in the assessment of patients to determine the level & degree of diagnostic & therapeutic intervention.APACHE II total score consists of three subheadings: acute physiology score, age and chronic health assessment; the highest value is 71. Mortality is 25% when the total score is 25, and increases to 80% when the total score is 35 and above.
Chelsea Critical Care Physical Assessment Tool (CPAx) | 3 days
  İt is a test used on male and female patients in the intensive care unit (ICU) to assess physical and respiratory function impairments and morbidity.
Body temperature | 3 days
  The average normal body temperature is generally accepted as 37°C. Some studies have shown that the "normal" body temperature can have a wide range, from 36.1°C to 37.2°C
Blood pressure | 3 days
  Normal blood pressure for most adults is defined as a systolic pressure of less than 120 and a diastolic pressure of less than 80. Elevated blood pressure is defined as a systolic pressure between 120 and 129 with a diastolic pressure of less than 80.
Respiratory rate | 3 days
  The normal range of breathing rate per minute in an average adult, for a person at rest, is 12 - 20 breaths per minute. Any person having a breathing rate under 12 or over 25 is considered to be breathing abnormally.
Pulse rate | 3 days
  The normal pulse for healthy adults ranges from 60 to 100 beats per minute. The pulse rate may fluctuate and increase with exercise, illness, injury, and emotions.
The Physical Function in ICU Test | 3 days
  The PFIT-s is a battery outcome measure involving four components: sit to stand assistance, marching on the spot cadence, shoulder flexor and knee extensor strength.
Hand Strength | 3 days
  Hand muscle strength will be measured with a jamar device
Modified Borg Dyspnea Scale | 3 days
  It is a categorical scale with a score from 0 to 10, where 0 represents normal breathing and 10 represents maximum dyspnea.
Pa02 | 3 days
  It is the partial pressure of oxygen in arterial blood. It is used to evaluate oxygenation.Normal values are 80-100 mmHg.
PaC02 | 3 days
  It is the partial pressure of carbon dioxide in arterial blood. It is an indicator of alveolar ventilation. Normal values are 35-45 mmHg.
HCO3 | 3 days
  It is the serum concentration of bicarbonate ion. It is an important buffer in the blood and is used to evaluate the metabolic component of acid-base balance. Standard bicarbonate: It is the bicarbonate value that should be present in the blood under standard conditions (37°C temperature and 40 mmHg PCO2). Normally it is 22-26 mEq/L.
Ph | 3 days
  It is used to determine the H+ status of the blood. It shows that the patient is in acidosis or alkalosis, but it is not possible to understand the type by pH. Normal values are 7.35-7.45.
Confusion Assessment Method for the ICU | 3 days
  The Confusion Assessment Method for the Intensive Care Unit (CAM-ICU) is a tool used to assess delirium among patients in the intensive care unit. The CAM-ICU assesses for the four features of delirium:Feature 1 is an acute change in mental status or a fluctuating mental status, Feature 2, is inattention, Feature 3,is altered level of consciousness and Feature 4, is disorganized thinking.
  patients in the intensive care unit

CONTACTS AND LOCATIONS:
Overall Officials: Yasemin Çırak, Prof Dr., Study Director — İstinye University

IPD SHARING:
Plan to Share IPD: No
Study Protocol, Statistical Analysis Plan (SAP), Informed Consent Form (ICF), Clinical Study Report (CSR) might be considered to be shared with clinicians studying in the same field one year after the publication of the study

REFERENCES:
- [Background] Berger D, Bloechlinger S, von Haehling S, Doehner W, Takala J, Z'Graggen WJ, Schefold JC. Dysfunction of respiratory muscles in critically ill patients on the intensive care unit. J Cachexia Sarcopenia Muscle. 2016 Sep;7(4):403-12. doi: 10.1002/jcsm.12108. Epub 2016 Mar 9. PMID 27030815
- [Background] Makhabah DN, Martino F, Ambrosino N. Peri-operative physiotherapy. Multidiscip Respir Med. 2013 Jan 23;8(1):4. doi: 10.1186/2049-6958-8-4. PMID 23343253
- [Background] Yousefnia-Darzi F, Hasavari F, Khaleghdoost T, Kazemnezhad-Leyli E, Khalili M. Effects of thoracic squeezing on airway secretion removal in mechanically ventilated patients. Iran J Nurs Midwifery Res. 2016 May-Jun;21(3):337-42. doi: 10.4103/1735-9066.180374. PMID 27186214
- [Background] Kalanuria AA, Ziai W, Mirski M. Ventilator-associated pneumonia in the ICU. Crit Care. 2014 Mar 18;18(2):208. doi: 10.1186/cc13775. No abstract available. PMID 25029020
- [Background] Ratnovsky A, Elad D, Halpern P. Mechanics of respiratory muscles. Respir Physiol Neurobiol. 2008 Nov 30;163(1-3):82-9. doi: 10.1016/j.resp.2008.04.019. Epub 2008 May 15. PMID 18583200
- [Background] Castro-Avila AC, Seron P, Fan E, Gaete M, Mickan S. Effect of Early Rehabilitation during Intensive Care Unit Stay on Functional Status: Systematic Review and Meta-Analysis. PLoS One. 2015 Jul 1;10(7):e0130722. doi: 10.1371/journal.pone.0130722. eCollection 2015. PMID 26132803
- [Background] Parker A, Sricharoenchai T, Needham DM. Early Rehabilitation in the Intensive Care Unit: Preventing Physical and Mental Health Impairments. Curr Phys Med Rehabil Rep. 2013 Dec;1(4):307-314. doi: 10.1007/s40141-013-0027-9. PMID 24436844
- [Background] Morris D, Jones D, Ryan H, Ryan CG. The clinical effects of Kinesio(R) Tex taping: A systematic review. Physiother Theory Pract. 2013 May;29(4):259-70. doi: 10.3109/09593985.2012.731675. Epub 2012 Oct 22. PMID 23088702
- [Background] Jang MH, Shin MJ, Shin YB. Pulmonary and Physical Rehabilitation in Critically Ill Patients. Acute Crit Care. 2019 Feb;34(1):1-13. doi: 10.4266/acc.2019.00444. Epub 2019 Feb 28. PMID 31723900
- [Background] Zeng R, Tian K, Xiao Z. Effectiveness of thoracic kinesio taping on respiratory function and muscle strength in patients with chronic obstructive pulmonary disease: A protocol of randomized, double-blind placebo-controlled trial. Medicine (Baltimore). 2021 Apr 9;100(14):e25269. doi: 10.1097/MD.0000000000025269. PMID 33832089
- [Background] Denehy L, de Morton NA, Skinner EH, Edbrooke L, Haines K, Warrillow S, Berney S. A physical function test for use in the intensive care unit: validity, responsiveness, and predictive utility of the physical function ICU test (scored). Phys Ther. 2013 Dec;93(12):1636-45. doi: 10.2522/ptj.20120310. Epub 2013 Jul 25. PMID 23886842
- [Background] Corner EJ, Wood H, Englebretsen C, Thomas A, Grant RL, Nikoletou D, Soni N. The Chelsea critical care physical assessment tool (CPAx): validation of an innovative new tool to measure physical morbidity in the general adult critical care population; an observational proof-of-concept pilot study. Physiotherapy. 2013 Mar;99(1):33-41. doi: 10.1016/j.physio.2012.01.003. Epub 2012 Mar 30. PMID 23219649